CLINICAL TRIAL: NCT00384267
Title: Congenital and Neonatal Malaria in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Other Study IDs: 05-0119
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2008-09

CONDITIONS: Malaria
Keywords: malaria, infants, preterm babies, neonates, Mali
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood

GROUPS / COHORTS (1):
- Neonates: Inpatient

SUMMARY:
This study will look at blood samples taken from 300 preterm babies and newborns admitted for inpatient care at Hopital Gabriel Toure in Bamako, Mali, and to gather information that will help the investigators verify the role of malaria in illness of very small babies. Blood samples will be taken from the mothers so that the investigators can find out if they have a malaria infection and how their body fights malaria. The investigators will also determine whether the mother and newborn baby are infected with the same malaria parasite. The information from this study may be used to improve malaria treatment in very small babies. Mothers and babies whose blood is tested will receive treatment for malaria as recommended by the National Malaria Control Program (NCMP).

DETAILED DESCRIPTION:
The purpose of this cross-sectional study is to determine the rate of congenital and acquired malaria in inpatient neonates at a tertiary pediatric hospital in Bamako, Mali. The primary study endpoint will be the number of infants with malaria infection as detected by the positivity of one of the three malaria diagnosis assays. The secondary study endpoints will be: (1) the rate of congenital malaria, (2) the rate of acquired malaria, (3) the prevalence of antimalarial antibodies in neonates, and (4) the prevalence of specific hemoglobin types in the study population. Neonates of both sexes who weigh at least 2000g, are 0 - 28 days old, and are referred to the Unit of Reanimation and Neonatology of Hopital Gabriel Toure in Bamako, Mali, for inpatient care are eligible for enrollment in this two-year study. After informed parental consent is obtained, approximately 2 ml of venous blood will be collected for malaria diagnosis by OptiMal test, microscopy and polymerase chain reaction (PCR). If in the clinician's judgment drawing blood is not feasible, a small blood sample will be obtained by heel prick from the infants and tested for the presence of malaria parasites. If any of the three infant malaria tests is positive, parenteral quinine will be administered as per the National Malaria Control Program (NMCP) treatment guidelines. If malaria is detected in mothers, standard malaria therapy will be administered according to the National Malaria Control Program (NMCP) treatment guidelines. Blood will be obtained from mothers for molecular diagnosis of malaria infection and characterization of the genetic profile of mother's malaria infections.

ELIGIBILITY:
Inclusion Criteria: Neonates: 1) Preterm born before 37 weeks of pregnancy admitted for inpatient care at HGT or Neonates aged between 0 - 28 days admitted for inpatient care at HGT 2) Admission weight more than 2000 grams 3) Parental informed consent obtained and signed for infant participation Criteria for Mothers: - Consenting mother of an enrolled infant Exclusion Criteria: Neonates: 1) Outpatient infant 2) Infant weighing less than 2000g 3) Infants presenting the following symptoms of critical condition: bradycardy, gasp, severely altered general condition 4) Presence of severe anemia 5) Infants who are judged by the study physicians to be unfit for enrollment for any reason 6) Informed consent denied Criteria for Mothers: 1) Mothers with severe malaria (2) 2) Mothers with an acute severe disease 3) Mothers who are judged by the study physician to be unfit for enrollment for any reason 4) Informed consent denied

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cross-sectional analysis of 300 inpatient neonates of both sexes who weigh at least 2000g, are 0 - 28 days old and are referred to the Unit of Reanimation and Neonatology of Hopital Gabriel Toure, Bamako, Mali
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
# of neonates with malaria infection | Immediately upon entry

SECONDARY OUTCOMES:
The rate of acquired malaria | Immediately upon entry
Prevalence of antimalarial antibodies in neonates | Immediately upon entry
The rate of congenital malaria | Immediately upon entry
Prevalence of specific hemoglobin types in study population | Immediately upon entry

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Gabriel Toure, Bamako, Mali